CLINICAL TRIAL: NCT04333745
Title: Influence of Obesity on Oxalate Metabolism and Handling in Calcium Oxalate Stone Formers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Dean Assimos, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB300004693-OHM; P20DK119788 (NIH); UAB (Other: UAB)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Kidney Stone
Keywords: oxalate; kidney stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Controlled Dietary Study (Experimental): Participants will consume the controlled diet for five days. After one day on the diet, subjects will provide three 24-hour urine collections. On the last dayof the diet, subjects will come in a fasted state to ingest a small amount of carbon-13 oxalate and sucralose, with hourly urine collections and blood samples being taken before and after the ingestion.
  Interventions: Other: Controlled Diet; Dietary Supplement: Carbon-13 Oxalate and Sucralose Ingestion

INTERVENTIONS:
Other: Controlled Diet — Participant will consume a controlled low oxalate diet for five days
Dietary Supplement: Carbon-13 Oxalate and Sucralose Ingestion — Subjects will ingest a small amount of carbon-13 oxalate and sucralose, dissolved in water.

SUMMARY:
The primary goals of this study are to determine the contribution of dietary oxalate absorption, renal oxalate handling, and endogenous oxalate synthesis to urinary oxalate excretion in normal Body Mass Index (BMI) and obese calcium oxalate kidney stone formers.

ELIGIBILITY:
Inclusion Criteria:

* Normal Body Mass Index (≥ 18.5 to < 25); Obese Body Mass Index (≥ 30 to ≤ 45)
* Able to provide informed consent
* Willingness to consume controlled diet
* Composition of most recent stone > 50% calcium oxalate, no uric acid component
* First time or recurrent calcium oxalate stone former
* 24-hour urine collections with creatinine values within 20% of appropriate ratio of creatinine (mg)/body weight (kg) for gender, and with creatinine values that are consistent between collections (within 20% of each other)
* Willingness to stop supplements [vitamins, Ca (citrate or carbonate) and other minerals, herbal supplements, nutritional aids, probiotics] for 14 days before start and during study
* Willingness to not undertake vigorous exercise during the controlled dietary study
* Normal fasting blood Comprehensive Metabolic Panel
* Hemoglobin A1c < 6.5%
* No food allergies or intolerance to any of the food in study menus
* Permitted/willing to discontinue medications for kidney stone prevention, including thiazides, allopurinol, and febuxostat and citrate preparations, for 14 days before start and during the studies. They will be instructed to restart these medications at the conclusion of the study

Exclusion Criteria:

* Diabetes
* Abnormal fasting comprehensive metabolic panel (CMP)
* Hemoglobin A1c (HbA1c) result ≥ 6.5%
* Gout
* Estimated Glomerular Filtration Rate (eGFR) <60 ml/min/1.73m^2
* Primary hyperoxaluria
* Cystic fibrosis
* Cystinuria
* Uric acid stone former
* Utilization of immunosuppressive medication
* Nephrotic syndrome
* Enteric hyperoxaluria
* Gastrointestinal disorder that could impact oxalate transport
* Sarcoidosis
* Uncontrolled hypertension
* Renal tubular acidosis
* Primary hyperparathyroidism
* Liver disease
* Neurogenic bladder
* Urinary diversion
* Chronic diarrhea
* Bariatric surgery
* Active malignancy or treatment for malignancy within 12 months prior to screening
* Pregnancy
* Breast feeding/nursing
* Females of child bearing age who are not able to use an effective method of birth control during the study
* Mental/medical condition that is likely to impede successful study completion
* Illness including flu / common cold / fever 14 days before study and during study
* Diarrhea or other abnormal gastrointestinal event (e.g. abnormal bowel movements) 14 days before study or during study
* Antibiotic use within last 6 months (based on recommendations of the NIH Human Microbiome Project, Protocol A)
* Inability or unwillingness to undergo MRI

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Oxalate Excretion | Baseline through Day 5
  Urinary oxalate excretion from urine samples will be measured as mg/day

CONTACTS AND LOCATIONS:
Overall Officials: Dean Assimos, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Texas Southwestern Medical Center, Dallas, Texas